CLINICAL TRIAL: NCT01699971
Title: Randomized Controlled Study Comparing Three Different Techniques for Open
Brief Title: Randomized Controlled Study Comparing Three Different Techniques for Open Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Thorell, Assoc prof, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006/672-31/4
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lichtenstein (Active Comparator): Hernia repair with lichtenstein propylene mesh
  Interventions: Procedure: Hernia repair

INTERVENTIONS:
Procedure: Hernia repair — Hernia repair admodum Lichtenstein with polypropylene mesh
Procedure: Hernia repair — Hernia repair with Ultra Pro Hernia System (UHS)
Procedure: Hernia repair — Hernia repair with Prolene Hernia System(PHS)

SUMMARY:
The primary aim is to evaluate if PSH and/or ultrapro mesch reduces chronic groin pain postoperatively compared to lichtenstein mesh. The second aim is to evaluate quality of life, recovery from surgery and frequency of recurrencies in the three groups

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* unilateral primary hernia
* open surgery

Exclusion Criteria:

* Recurrent Hernia
* Bilateral Hernia
* laparoscopic surgery
* Female

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-10; Primary Completion 2009-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
postoperatively pain | Postoperative 36 month
  Visual analog scale (VAS)

SECONDARY OUTCOMES:
Quality of life | 36 month postoperative
  SF36
frequency of recurrencies | postopertive 36 month
  check patients journal

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, Assoc Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Ersta Hospital, Stockholm, Sweden